CLINICAL TRIAL: NCT00261066
Title: A Prospective Database for Orthopaedic Surgery
Brief Title: Outcome Following Orthopaedic Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: OHREB 2003209-01H
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Osteoarthritis of Knee
Keywords: Functional outcome; Orthopaedic surgery
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By investigating the long-term functional status of patients who have undergone various types of orthopaedic surgery we will have a basis for devising guidelines for future patients and surgeons.

DETAILED DESCRIPTION:
The purpose of this database is to explore the long term outcome and functional status of patients undergoing various types of orthopaedic surgery. These data will yield a valuable database that can be used to address future research questions. For example, there are three common surgical treatments for medial osteoarthritis of the knee: tibial osteotomy, Oxford partial knee replacement, or total knee replacement. No clear guidelines exist regarding which treatment options are optimal for which patients. By gathering functional data from patients who have undergone these treatments, we will have a basis for devising such guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are scheduled to undergo orthopaedic surgery are eligible to be included in the database.

Exclusion Criteria:

* Those patients who do not meet the above inclusion criteria will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to undergo orthopaedic surgery at The Ottawa Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 8439 (Actual)
Dates: Start 2003-05-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Koos | 10y
  baseline,1y-2y-5y-7y10y

SECONDARY OUTCOMES:
ShortForm-12 | 10Years
  baseline,1y-2y-5y-7y10y
Tegner-ulca | 10Years
  baseline,1y-2y-5y-7y10y

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Dervin, MD, Principal Investigator — OHRI
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided